CLINICAL TRIAL: NCT03129412
Title: The Clinical Curative Efficacy and Side Effect of Oligo-metastases Nasopharyngeal Carcinoma Patients Received Radical Radiation for Primary Tumors and Treatments for Metastatic Lesions
Brief Title: Oligo-metastases NPC Patients Received Radiation for Primary Tumors and Treatments for Metastatic Lesions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-Oligo-M
Record Dates: First submitted 2017-04-12; First posted 2017-04-26 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Cancer; Neoplasm Metastasis
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): 4-6 cycles chemotherapy and radical radiotherapy for primary tumors were given. Appropriate treatments for olio-metastatic lesions will assigned to those who got PR,SD after chemotherapy.
  Interventions: Radiation: radical radiotherapy

INTERVENTIONS:
Radiation: radical radiotherapy — radical radiotherapy for primary tumors were given. Appropriate treatments for olio-metastatic lesions will be assigned to those who got PR,SD after chemotherapy.

SUMMARY:
Oligo-metastases NPC patients received radiation for primary tumors and treatments for metastatic lesions.

DETAILED DESCRIPTION:
The patients enrolled will received 4-6 cycles chemotherapy at first.Then, radical radiotherapy for nasopharyngeal tumors and local treatments for oligometastatic lesions will assigned to those patients. The efficacy and side-effect will be evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically conformed initial non-keratinizing squamous carcinoma in nasopharynx.
2. Clinical stages,T1-4N0-3M1，IVc(AJCC 2010).
3. The metastatic lesions ≤5 and metastatic organs ≤2
4. Karnofsky scores >70
5. Normal hemodynamic indices before the recruitment (including white blood cell count>4.0×109/L, neutrophil count>1.5×109/L, platelet count >100×109/L, hemoglobin≥90g/l, normal liver/kidney function).
6. Informed consent signed.

Exclusion Criteria:

1. Histologically conformed initial keratinizing carcinoma or others.
2. The metastatic lesions >5 or metastatic organs >2.
3. Any severe complications contraindicated chemotherapy or radiotherapy.
4. History of malignant tumors.
5. Pregnant or nursing women.
6. History of radiotherapy or chemotherpy in head and neck regions.
7. Patients refused the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2023-04-23 (Estimated); Study Completion 2025-04-23 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Events of death caused by any reasons

SECONDARY OUTCOMES:
Progress free survival | From date of diagnosis until the date of first documented progression, assessed up to 36 months
  adverse event including death, recurrence and metastases.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No